CLINICAL TRIAL: NCT04705545
Title: Anchorage Reinforcement in Bimaxillary Proclination Cases - a 3-arm Randomised Controlled Trial
Brief Title: Anchorage Reinforcement in Bimaxillary Proclination Cases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Kumeran Mohan, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UM_ORTHO_KM001
Record Dates: First submitted 2020-11-29; First posted 2021-01-12 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Bimaxillary Proclination
Keywords: bimaxillary proclination; anchorage; soft tissue changes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- molar block (No Intervention): No additional anchorage reinforcements besides the banding first and second molar with and tying them together at the buccal tubes (also known as molar block)
- TPA group (Experimental): Bands are selected and an alginate impression taken over the bands. The impression will be sent to the lab for the construction of a transpalatal archwire on a 1.0 mm stainless steel wire connecting the upper permanent first molar, with a U loop pointing posteriorly, soldered to the palatal side of the molar bands. The appliance will be fitted a week later. Molar bands will be fitted to the permanent second molar on the same appointment, with a ligature wire tying the first molar band together at the buccal tubes. The resulting anchorage reinforcement is a molar block with a transpalatal archwire.
  Interventions: Device: transpalatal arch group
- Nance button group (Experimental): Bands are selected and an alginate impression taken over the bands. Bands are replaced on the tooth and an alginate impression taken over the bands. The impression will be sent to the lab for the construction of a transpalatal archwire on a 1.0 mm stainless steel wire connecting the upper permanent first molar, with a Nance button incorporated in the middle of the wire, soldered to the palatal side of the molar bands. The appliance will be fitted a week later. Molar bands will be fitted to the permanent second molar on the same appointment, with a ligature wire tying the first molar band together at the buccal tubes. The resulting anchorage reinforcement is a molar block with a Nance button
  Interventions: Device: Nance button

INTERVENTIONS:
Device: transpalatal arch group — transpalatal arch is a 1.0 mm stainless steel wire connecting the upper permanent first molar, with a U loop pointing posteriorly, soldered to the palatal side of the molar bands.
  Other Names: TPA
  Arms: TPA group
Device: Nance button — Nance button is a 1.0mm stainless steel wire connecting the upper permanent first molar, with a Nance button incorporated in the middle of the wire, soldered to the palatal side of the molar bands
  Arms: Nance button group

SUMMARY:
Bimaxillary protrusion are common in Malaysia due to the prevalence in the two biggest races (Malay and Chinese). However, evidence for treatment methods and outcomes for bimaxillary protrusion patients are scarce. The need for high anchorage in bimaxillary protrusion cases also makes them perfect candidates for a study on the effectiveness of different anchorage methods commonly used in treatment of bimaxillary protrusion cases. The soft tissue outcomes from the use of these different methods are also our area of interest. Hence, the investigators aim is to prove that molar block anchorage similarly effective and has the same outcome as using other conventional auxiliary anchorage such as TPA and Nance button in treating patients with bimaxillary protrusion.

DETAILED DESCRIPTION:
Bimaxillary proclination is common in Malaysia especially among Malay, Chinese and possibly the Malaysian Aborigines. Treatment commonly constitutes extraction of upper and lower first permanent premolars with maximum anchorage requirement. Various anchorage device exists, but conventional devices such as Nance button, transpalatal arch and molar blocks are still commonly used to good effect in treatment of bimaxillary proclination. A comparison of these commonly used conventional anchorage devices (molar block, transpalatal arch, Nance button), especially in treating bimaxillary proclination cases, surprisingly has not been done.

Soft tissue changes also occur in bimaxillary proclination. However, changes in the soft tissue profile using these conventional anchorage devices do not exist, as evidence shows that anchorage devices can affect soft tissue outcomes

Hence, the investigators aim to investigate compare the effectiveness and soft tissue changes of using just molar blocks, molar blocks with transpalatal arch and molar blocks with Nance button.

This study will be done as a 3-arm parallel randomised controlled trial. The allocation ration is set at 1:1:1. This study will adhere to the PICO and CONSORT guidelines, and will be registered with the clinical.org website.

Sample size calculation was conducted using G Power 3.9.1.4. The standard deviation of the movement of maxillary permanent first molar was estimated at 2.2 mm. The mean difference of 1.00 mm was considered the smallest important difference to be detected, which was also used as the effect size. In order to detect the difference of 1.00 mm with a power of 0.80 (80%) and an alpha of 0.05, accounting for a 20% dropout, the total sample size required is 15, which will be randomised into 3 groups (5 Nance group, 5 TPA group and 5 molar block group).

Each patient will be randomised by the following protocol. A simple stratified randomisation method is done with gender as the stratification factor, using Sealed Envelope Ltd. 2019. Each allocation is written on a paper, which will be folded twice (to reduce bias), placed in separate opaque envelopes and sealed. The envelopes will be coded by gender using stickers and numbered in sequence. Each gender will have their own sequence of numbers (male: 1-16, female: 1-17). The envelopes will be stored in a locked drawer in the Orthodontic Dental Clinic.

Eligible patients are then screened from the orthodontic waiting list by three operator clinicians according to the inclusion and exclusion criteria set. Patients identified will be given an explanation on the trial and will be invited to take part. Upon receiving informed consent from patients, the envelope will be allocated to patients according to the number sequence.

Full orthodontic examination, records taking (pre-treatment radiograph (cephalometric radiographs, panoramic radiographs, and other necessary additional periapical radiographs), photographs and study models) and treatment planning will be done. The pre-treatment study model will be labelled as T0.

The following treatment protocol is then followed:

Group A: No additional anchorage reinforcements besides the banding first and second molar with and tying them together at the buccal tubes (also known as molar block).

Group B: Bands are selected and an alginate impression taken over the bands. The impression will be sent to the lab for the construction of a transpalatal archwire on a 1.0 mm stainless steel wire connecting the upper permanent first molar, with a U loop pointing posteriorly, soldered to the palatal side of the molar bands. The appliance will be fitted a week later. Molar bands will be fitted to the permanent second molar on the same appointment, with a ligature wire tying the first molar band together at the buccal tubes. The resulting anchorage reinforcement is a molar block with a transpalatal archwire.

Group C: Bands are selected and an alginate impression taken over the bands. Bands are replaced on the tooth and an alginate impression taken over the bands. The impression will be sent to the lab for the construction of a transpalatal archwire on a 1.0 mm stainless steel wire connecting the upper permanent first molar, with a Nance button incorporated in the middle of the wire, soldered to the palatal side of the molar bands. The appliance will be fitted a week later. Molar bands will be fitted to the permanent second molar on the same appointment, with a ligature wire tying the first molar band together at the buccal tubes. The resulting anchorage reinforcement is a molar block with a Nance button

Next, patients will undergo planned extraction of upper and lower permanent first premolars.

Treatment is started with alignment and levelling using preadjusted Edgewise fixed appliances (Gemini McLaughlin, Bennett, Trevisi (MBT) Twin Bracket 5x5 [3M Unitek, Monrovia, CA, USA] prescription; 0.022-in slot size) following a straight wire concept on the upper and lower arches. The wire sequence used were as follows i. 0.016-in heat activated Nickel Titanium [3M Unitek], ii. 0.018 x 0.025-in heat activated Nickel Titanium [3M Unitek], iii. 0.019 x 0.025-in stainless steel [3M Unitek]).

At this point, a snap impression is taken (T1).

Before impression taking, a marking is done on the upper first molar buccal cusps with indelible ink to mark the position of the molar band. The molar bands (with or without the Nance button or TPA) will be removed. A satisfactory upper arch snap impression is taken. The molar bands (with or without the anchorage reinforcement device) are recemented on the teeth using the mark on the buccal cusp to improve accuracy and reduce bias.

Next, space closure is done using intramaxillary traction mechanics using primarily Nickel Titanium alloy closed coil springs, due to their consistent and efficient force delivery compared to elastomeric chains. The completion of space closure will be assumed when all spaces are closed. At this point, the auxiliary anchorage reinforcements are removed (Nance button or TPA), leaving just the molar blocks (molar band on first and second permanent molars). A snap impression will be taken at completion of space closure (T2). A cephalometric radiograph is also taken. Treatment is continued and completed as planned for every patient involved in the study.

The models (T0, T1 and T2) will be sent to the 3D Gens Lab to be scanned, to obtain digital 3-dimensional models in STL format. Superimposition will be done by Mimics software which allows 3D superimposition and measurements to be done. We will use a designated stable area on the palate, which allows measurements in all three planes. In our study, we will be using the 'mushroom area' of the palate, which is a stable structure commonly used for superimposition, even in growing patients. It is also an area which is easier to designate due to the area covered. The area of the palate covered includes:

* anteriorly: the medial 2/3 of the third rugae anteriorly
* laterally: two lines parallel to the midpalatal suture laterally
* posteriorly: 5 mm from the third rugae posteriorly
* extending to the level of an imaginary line connecting the lingual grooves of the 1st permanent molars.

The treatment and impressions will be done by 2 operators. The following superimposition & measurement of the 3-dimensional dental casts will be done by a single researcher in all 3 planes. Finally, before the digital model superimposition and measurements are done, 10 random models will be superimposed and measured first. The process will be repeated in 2 weeks for an inter-class correlation coefficient (ICC) to assess intra-rater reliability of the superimposition and measurement procedure.

Due to the nature of this study, no blinding will be done on the patient or the treating operator as it would not be possible. Blinding will be done during the data collection and analysis stage by coding every patient before sending the models to the lab for data processing and collection. A single researcher will be handling all the data.

The statistical analysis for this study will be done using SPSS statistics version 23 [IBM, Illinois, USA]. The raw data will first be tested for normal distribution, followed by descriptive statistics using a demographic characteristics chart. Next, an analysis of covariance (ANCOVA), with gender as a stratifying factor will be done, where probabilities less than 5% (P < 0.05) will be considered significant. Data will also be analysed on an intention-to-treat basis, to take into account any unsuccessful or dropout cases. An ICC will also be done to assess the intra-rater reliability in superimposing and measurements.

ELIGIBILITY:
Inclusion Criteria:

Patients with:

* a need to correct bimaxillary proclination
* age of 16 years old and above
* a need for extraction of the permanent first premolars
* mild space requirement (less than 4mm), no crowding or spaced dentition
* good oral hygiene

Exclusion Criteria:

Patient with

* hypodontia
* history of orthodontic treatment or extractions (except third molars)
* congenital oral-maxillofacial deformities such as cleft lip and palate
* syndromic diseases
* orthognathic treatment need
* poor dental health precluding orthodontic treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
molar movement | 24 months
  Three plane movement of the maxillary permanent first molar in terms of anchorage loss (in mm)
Soft tissue cephalometric changes (angle) | 24 months
  Nasolabial angle, H angle and facial convexity angle
Soft tissue cephalometric changes (degrees) | 24 months
  E line, labiomental sulcus depth, upper lip length, lip protuberance

SECONDARY OUTCOMES:
Duration of treatment visits (minutes) | 24 months
  Duration of treatment visits (T0 - T2)
Number of treatment visits (days) | 24 months
  Number of treatment visits (T0 - T2)
Hard tissue cephalometric changes (degrees) | 24 months
  S-N-A point angle, S-N-B point angle, A-N-B point angle, Maxillary-Mandibular Plane angle

CONTACTS AND LOCATIONS:
Overall Officials: Siti A Othman, MOrthRCSEd, Study Director — Faculty of Dentistry, University Malaya
Locations (1):
- Faculty of Dentistry, University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alqahtani ND, Alshammari R, Almoammar K, Almosa N, Almahdy A, Albarakati SF. Post-orthodontic cephalometric variations in bimaxillary protrusion cases managed by premolar extraction - A retrospective study. Niger J Clin Pract. 2019 Nov;22(11):1530-1538. doi: 10.4103/njcp.njcp_125_19. PMID 31719274
- [Background] Dixon V, Read MJ, O'Brien KD, Worthington HV, Mandall NA. A randomized clinical trial to compare three methods of orthodontic space closure. J Orthod. 2002 Mar;29(1):31-6. doi: 10.1093/ortho/29.1.31. PMID 11907307
- [Background] Samuels RH, Rudge SJ, Mair LH. A comparison of the rate of space closure using a nickel-titanium spring and an elastic module: a clinical study. Am J Orthod Dentofacial Orthop. 1993 May;103(5):464-7. doi: 10.1016/S0889-5406(05)81798-6. PMID 8480716
- [Background] Ganzer N, Feldmann I, Bondemark L. Anchorage reinforcement with miniscrews and molar blocks in adolescents: A randomized controlled trial. Am J Orthod Dentofacial Orthop. 2018 Dec;154(6):758-767. doi: 10.1016/j.ajodo.2018.07.011. PMID 30477773
- [Background] Solem RC, Marasco R, Guiterrez-Pulido L, Nielsen I, Kim SH, Nelson G. Three-dimensional soft-tissue and hard-tissue changes in the treatment of bimaxillary protrusion. Am J Orthod Dentofacial Orthop. 2013 Aug;144(2):218-28. doi: 10.1016/j.ajodo.2013.03.018. PMID 23910203
- [Background] Vasilakos G, Schilling R, Halazonetis D, Gkantidis N. Assessment of different techniques for 3D superimposition of serial digital maxillary dental casts on palatal structures. Sci Rep. 2017 Jul 19;7(1):5838. doi: 10.1038/s41598-017-06013-5. PMID 28724930